CLINICAL TRIAL: NCT05169762
Title: Feminizing Treatment in Transgender Women and Non-binary Persons BODY IDENTITY CLINIC - ESTROGEN
Brief Title: Feminizing Treatment in Transgender Women and Non-binary Persons
Acronym: BIC-Estrogen
Status: Recruiting | Type: Observational
Sponsor: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Marianne Andersen, Clinical professor, Odense University Hospital
Other Study IDs: BICTX03
Record Dates: First submitted 2021-09-19; First posted 2021-12-27 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Transgenderism
Keywords: gender affirming hormone treatment; estrogen; cardiovascular risk
MeSH Terms: conditions — Transsexualism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- transgender women: transgender women eligeble to start gender affirming hormone treatment
  Interventions: Other: standard treatment

INTERVENTIONS:
Other: standard treatment — starndard treatment for transgender women

SUMMARY:
Cohort study in 100 transgender women treated with gender affirming hormone treatment. Follow up affter 1year, 3 years, 5 years and 10 years, Outcomes regarding cardiovascular effects of hormone treatment.

DETAILED DESCRIPTION:
Cohort study in 100 transgender women treated with gender affirming hormone treatment. Follow up affter 1year, 3 years, 5 years and 10 years,

Outcomes:

Non-calcified and calcified plaque formation by contras coronary CT angiograms Heartfunction by ekko Cardiovaskular risk markers, f. eks. bp Markers of cardiovascular risk in blood and urine

ELIGIBILITY:
Inclusion Criteria:

* assigned male at birth and eligeble for gender affirming feminizing treatment

Exclusion Criteria:

none

-

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — assigned male at birth, identifiing as transgender women
Study Population: transgender women
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2035-09-01 (Estimated); Study Completion 2035-09-01 (Estimated)

PRIMARY OUTCOMES:
coronary plaque formation | 1 year
  mm3

CONTACTS AND LOCATIONS:
Overall Officials: Dorte Glintborg, Principal Investigator — Odense University Hospital
Locations (1):
- OdenseUH, Odense, Denmark

IPD SHARING:
Plan to Share IPD: No